CLINICAL TRIAL: NCT06731361
Title: Improving Medication Prescription in the contExt of Advance Care Planning for paTients Receiving Long Term nUrSing Home Care
Brief Title: Improved Prescribing for Older Nursing Home Patients
Acronym: IMPETUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Martin Smalbrugge, Principal investigator, professor of Medicine for Older People and chair of the Department of Medicine for Older People, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 839160003
Record Dates: First submitted 2024-08-14; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Nursing Home Residents; Older People; Prescribing; Advance Care Planning; Medication Reviews; Decision Making; Prescribing Practices
Keywords: limited life expectancy; ReNeWAL criteria (adjusted STOPP/START criteria); decision making involvement; appropriate prescribing; Cluster randomised trial; Educational intervention; Prescribing practices

STUDY DESIGN:
Intervention Model Description: Cluster randomised controlled trial with 2 arms: intervention and control. Ratio 1:1. 2 clusters start in september, 2 clusters start in october and 2 clusters start in november.
Masking Description: Not possible due to the type of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group, care as usual
- Educational intervention (Experimental): The clusters that fall into the experimental arm receive the educational intervention: they receive an in-house training in combination with supporting tools, educational materials and intervision moments.
  Interventions: Combination Product: Systematic multidisciplinary medication review + ACP (SMMR+)

INTERVENTIONS:
Combination Product: Systematic multidisciplinary medication review + ACP (SMMR+) — The intervention is a training in medication assessment. The goal is to align prescription with the treatment goals of nursing home patients which are set in advance care planning conversations. The training consists of 2 components:
  1. Medication assessment with the use of the ReNeWAL criteria (adjusted STOPP/START criteria, tailored to nursing home patients with a limited life expectancy)
  2. Advance care planning component. Discussing medication in line with the treatment goals set in advance care planning conversations.
  Healthcare professionals receive the training in combination with supporting tools (pocket card) and educational material (the ReNeWAL criteria and PowerPoint slides of the training if requested). Also, intervision moments are planned.
  Other Names: ReNeWAL criteria; Pocket card
  Arms: Educational intervention

SUMMARY:
Research aim:

To investigate the effect of training health care professionals in medication assessments on the medication use of nursing home residents with a limited life expectancy (< 1.5-2 years).

The core of the training is to tailor medication use to (palliative) treatment goals of nursing home residents.

Design:

A cluster randomized controlled trial on long term care wards in nursing homes, with the nursing home care organisations as unit of randomisation. The investigators intent to include 6 organisations and 450 nursing home patients. The research starts in september and lasts 1 year and 3 months. Eligible patients are nursing home patients of 65 years and older with a limited life expectancy (< 1.5-2 year) of long term care wards.

Intervention:

The intervention includes a method in which healthcare professionals (medical practitioner, pharmacist and care worker) are trained to tailor medication to the (palliative) treatment goals of nursing home patients with a limited life expectancy. The training consists of 2 components: 1) medication assessment, and 2) advance care planning (ACP). In the intervention group, healthcare professionals receive the training in combination with supporting tools and educational materials, in the control group care continues as normal. The allocation ratio for control and intervention groups is 1:1. A process evaluation will take place simultaneously with the intervention study. Data collection takes place before the start of the intervention (T0), after 6 months (T1) and after 12 months (T2).

Outcome measures:

The primary outcome measure is potential under- and over-treatment with medication. The secondary outcome measure is experienced involvement in decision-making (measured with a short questionnaire based on the revised PATD (patients' attitude towards deprescribing)). Tertiary outcome measures are: quality of life, deaths, falls, hospital admissions/acute first aid referrals and pain.

Discussion:

The intervention is expected to result in a decrease in chronic and preventive medication prescriptions, an increase in medication for symptom treatment and more involvement (and satisfaction) of the nursing home resident in decision-making, without adverse effects.

DETAILED DESCRIPTION:
Additional information on the method:

We included 2 nursinghome organizations in september, 2 in october, and 3 in november.

ELIGIBILITY:
Inclusion Criteria:

Nursing home patients:

* Age 65years and above
* Living at long term care wards in nursing homes
* Living at a long term care ward for at least 4 weeks before start of the study

Exclusion Criteria:

* Temporary nursing home patients (i.e. geriatric rehabilitation or end-of-life/hospice care)
* Life expectancy < 4 weeks
* Life expectancy clearly > 1.5 - 2 years (i.e. patients with Huntingtons disease)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Potential under- and overprescribing | at baseline - 6 months - 12 months
  Potential under- and overprescribing

SECONDARY OUTCOMES:
Experienced involvement in decision-making | At baseline and 2-4 weeks after the medication review
  Experienced involvement in decision-making measured with a questionnaire

OTHER OUTCOMES:
QOL (Quality of life) | at baseline - 6 months - 12 months
  Quality of life measured with the EuroQol questionnaire (EQ-5D)
Social wellbeing | at baseline - 6 months - 12 months
  Measured with Revised index for social engagement (RISE) questionnaire
Adverse outcomes | at baseline - 6 months - 12 months
  Adverse outcomes, such as: deaths, falls, hospital admissions/acute referrals, measured over the previous 6 months. (Only for ' deaths' not possible at baseline.)
Pain assessment | at baseline - 6 months - 12 months
  measured with the pain items of the Resident Assessment Instrument for Long-term Care Facilities (RAI-LTCF) questionnaire
Process evaluation | Through 1 year and 3 months
  Qualitative and quantitative data

CONTACTS AND LOCATIONS:
Overall Officials: Martin Smalbrugge, Prof, Study Director — Amsterdam UMC, location VUmc, departement Medicine for Older People
Locations (7):
- Netherlands (7):
  - Zorggroep Apeldoorn, location Randerode, De Hofstede and De Windkanter, Apeldoorn, Gelderland
  - Zorggroep Noordwest-Veluwe, locaties Weideheem en de Arcade, Harderwijk, Gelderland
  - Cordaan, location Nieuw Vredenburgh, Amsterdam, North Holland
  - Amaris, Location Alporti and Rubina, Hilversum, North Holland
  - AxionContinu, location Isselwaerde and de Schutse, IJsselstein, Utrecht
  - Zorgspectrum, location de Plataan, Vianen, Utrecht
  - Dignis, location de Veldspaat, Groningen

IPD SHARING:
Plan to Share IPD: No